CLINICAL TRIAL: NCT01781585
Title: The Hemodynamic Effects During Sustained Low-efficiency Dialysis Versus Continuous Veno-venous Hemofiltration for Patients With Intracranial Hypertension in a Cross Over Study (NSARF)
Brief Title: The Hemodynamic Effects During Sustained Low-efficiency Dialysis Versus Continuous Veno-venous Hemofiltration for Patients With Intracranial Hypertension in a Cross Over Study
Acronym: NSARF
Status: Withdrawn | Type: Observational
Why Stopped: Inclusion criteria difficulties to receive the case, it is taken off the case to apply
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201107015RC
Record Dates: First submitted 2012-09-17; First posted 2013-02-01 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: End- Stage Renal Disease Patients
Keywords: Sustained low-efficiency dialysis;; Continuous venovenous hemofiltration;; hemodynamic stability,; Intracranial pressure
MeSH Terms: interventions — Renal Dialysis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- sustained low-efficiency dialysis: Patients were randomized to receive CVVH or SLED and the next day on the other.
  Interventions: Procedure: hemodialysis
- continuous veno-venous hemofiltration: Patients were randomized to receive CVVH or SLED and the next day on the other.
  Interventions: Procedure: hemodialysis

INTERVENTIONS:
Procedure: hemodialysis — Patients were randomized to receive CVVH or SLED and the next day on the other.

SUMMARY:
Hemodynamic instability occurs frequently during dialysis treatment and still remains as significant cause of patient mobility and mortality. Postoperative hemodynamic optimization has been proved to reduce morbidity in high-risk patients. Intracranial pressure increased can lead to further structural and functional impairment owing to its deleterious effect on the compromised microcirculation and metabolism. This study was to compare the intra-cerebral pressure (ICP) and hemodynamic parameters between the sustained low-efficiency dialysis (SLED) and continuous veno-venous hemofiltration (CVVH) in post- brain tramatic patients.

DETAILED DESCRIPTION:
Patients and Methods This study was based on a clinical cohort study of the renal failure patients in the database of the National Taiwan University Surgical ICU Acute Renal Failure (NSARF) Study Group17-21, with the approval of the Institutional Review Board of the National Taiwan University Hospital (201107015RC).

Study protocol

The inclusion criteria were end stage renal disease (ESRD) patients with increased ICP status post ICP monitor insertion. We started the study after the hemodynamic stable and acceptable ICP less than 20mmHg22. The ESRD patients with active brain hemorrhage, cardiac arrhythmia during dialysis, residual urine output, with inotropic equivalent more than 15 were excluded.

All the patients were ventilated in supine position in controlled-volume mode after stable from brain hemorrhage. During data collection, supportive therapies, ventilatory settings and vasopressor therapy were kept unchanged. Patients were randomized to receive CVVH or SLED and the next day on the other. The ICP monitor was equipped and the indwelling radial artery catheter connected to the FloTrac/Vigileo hemodynamic monitoring system and for whom the ultrafiltration rate was set around 1.0 kg/8hr to 1.5 kg/8hr according to fluid status. Ultrafiltration rate and sodium concentration were fixed during each session.

Clinical assessment The biochemical parameters were measured using the Toshiba TBA-200FR Clinical Chemistry Analyzer (Toshiba, Tochigi-Ken, Japan). When multiple daily measurements were performed, the data obtained closest to 8:00 AM were analyzed 23. The baseline hemodynamic was defined as average of two hours prior dialysis in each dialysis sessions.

ELIGIBILITY:
Inclusion Criteria:

* end-stage kidney disease with anuria status post ICP monitor insertion received

Exclusion Criteria:

* acute dialysis patients
* end-stage kidney disease with uria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The inclusion criteria were end stage renal disease (ESRD) patients with increased ICP status post ICP monitor insertion
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
hemodynamic stability during dialysis | 2days
  Cardiac output and stroke volume variation measurements and ICP measurement

SECONDARY OUTCOMES:
the difference between cardiovascular peptides, oxidative and inflammatory assays | 2 days
  the difference between cardiovascular peptides, oxidative and inflammatory assays

CONTACTS AND LOCATIONS:
Overall Officials: VinCent Wu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Daugirdas JT. Dialysis hypotension: a hemodynamic analysis. Kidney Int. 1991 Feb;39(2):233-46. doi: 10.1038/ki.1991.28. No abstract available. PMID 2002637
- [Background] Zager PG, Nikolic J, Brown RH, Campbell MA, Hunt WC, Peterson D, Van Stone J, Levey A, Meyer KB, Klag MJ, Johnson HK, Clark E, Sadler JH, Teredesai P. "U" curve association of blood pressure and mortality in hemodialysis patients. Medical Directors of Dialysis Clinic, Inc. Kidney Int. 1998 Aug;54(2):561-9. doi: 10.1046/j.1523-1755.1998.00005.x. PMID 9690224
- [Derived] Wu VC, Huang TM, Shiao CC, Lai CF, Tsai PR, Wang WJ, Huang HY, Wang KC, Ko WJ, Wu KD; NSARF Group. The hemodynamic effects during sustained low-efficiency dialysis versus continuous veno-venous hemofiltration for uremic patients with brain hemorrhage: a crossover study. J Neurosurg. 2013 Nov;119(5):1288-95. doi: 10.3171/2013.4.JNS122102. Epub 2013 May 24. PMID 23706048